CLINICAL TRIAL: NCT07292519
Title: Tirzepatide Combined With Cognitive-Behavioural Therapy (CBT) for Adults With Alcohol Use Disorder (AUD) and Overweight/Obesity (OOB)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Collaborators: The University of Sydney, Sydney, Australia (Unknown)
Responsible Party: Principal Investigator, Kirsten Morley BPsych MPH PhD, Professor, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X25-0171
Record Dates: First submitted 2025-12-01; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD); Overweight or Obese; Comorbidities and Coexisting Conditions
Keywords: Alcohol Use Disorder (AUD); Overweight or Obese; Concurrent Treatment of AUD and overweight/obesity; Tirzepatide; Phase II Double-blind RCT
MeSH Terms: conditions — Alcoholism; Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: Phase II, double blind, placebo-controlled RCT designed to assess the efficacy (on alcohol consumption, craving and cardiometabolic outcomes) and safety of tirzepatide for individuals with alcohol use disorder and overweight/obesity (AUD-OOB).
  Participants will receive 8 weekly doses of tirzepatide or placebo (from visit 2, week 1 to visit 9, week 8) administered sub-cutaneously combined with structured "Take Control" CBT sessions (from visit 2, week 1 to visit 10, week 8), followed by follow-up assessments.
Who Masked: Participant, Investigator
Masking Description: Randomisation will be carried out using a computer-generated list prepared by an independent biostatistician who is not involved in participant recruitment or assessment. The randomisation schedule will be securely uploaded to REDCap and accessible only to unblinded pharmacy staff responsible for study drug dispensing. Investigators enrolling participants will remain blinded and will not have access to the allocation list at any stage. Unblinding will only be permissible in the event of a medical emergency where knowledge of the participant's treatment assignment is essential to inform clinical care. Such unblinding will be conducted by the study pharmacist and must be documented and justified in the participant's trial record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide: subcutaneous administration of Tirzepatide plus CBT ("Take Control" program) (Experimental): 1 x Screening, Baseline Clinical Assessments, Neuroimaging (T0) and Psychophysiology, Randomisation (Visit 1, Week 0)
  From Dose 1 (Visit 2, week 1) to Dose 4 (Visit 5, week 4), with "Take Control" CBT module: 2.5mg Tirzepatide dose administration, and a 15-20 minutes computer-based CBT module.
  From Dose 5 (Visit 6 , week 5) to Dose 8 (Visit 9, week 8) with "Take Control" CBT module: 5.0mg dose administration (unless contraindicated by study physician), and a 15-20 minutes computer-based CBT module.
  Neuroimaging substudy (Visit 10, week 8): After the final medication and CBT module, participants complete final neuroimaging timepoint (T1).
  End-of-treatment (Visit 11, week 9 & Visit 12, week 12): One and four weeks after the last dose and neuroimaging, participants will complete psychophysiology assessments using the same tasks as baseline.
  Interventions: Drug: Tirzepatide; Behavioral: Take Control CBT Module
- Placebo: subcutaneous administration of placebo plus CBT ("Take Control" program) (Placebo Comparator): 1 x Screening, Baseline Clinical Assessments, Neuroimaging (T0) and Psychophysiology, Randomisation (Visit 1, Week 0)
  From Dose 1 (Visit 2, week 1) to Dose 4 (Visit 5, week 4), with "Take Control" CBT module: matched placebo dose administration OR matched placebo, and a 15-20 minutes computer-based CBT module.
  From Dose 5 (Visit 6 , week 5) to Dose 8 (Visit 9, week 8) with "Take Control" CBT module: matched placebo administration, and a 15-20 minutes computer-based CBT module.
  Neuroimaging substudy (Visit 10, week 8): After the final medication and CBT module, participants complete final neuroimaging timepoint (T1).
  End-of-treatment (Visit 11, week 9 & Visit 12, week 12): One and four weeks after the last dose and neuroimaging, participants will complete psychophysiology assessments using the same tasks as baseline.
  Interventions: Behavioral: Take Control CBT Module; Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Subcutaneous injection once weekly for 8 weeks: 2.5 mg/week initially for Weeks 1-4, then 5.0 mg/week for Weeks 5-8 (Dose escalation from 2.5 mg to 5.0 mg will occur at Week 5 unless the study physician advises continuation at the lower dose due to tolerability concerns. Delays or dose adjustments will be made per the physician's clinical judgment).
  Other Names: GLP-1/GIP receptor dual agonist
  Arms: Tirzepatide: subcutaneous administration of Tirzepatide plus CBT ("Take Control" program)
Behavioral: Take Control CBT Module — The Take Control intervention is a structured CBT intervention or manualised digital therapy designed to support alcohol reduction.
  Take Control will be completed using a computer interface with headphones in a private room. Participants will complete one module per week during treatment Weeks 1 to 8. Each module is approximately 30-45 minutes in length and will be completed independently by the participant under the supervision of a research assistant. Program content is fixed and self-paced, eliminating the need for fidelity monitoring of therapist behaviour.
  Take Control is an evidence-informed cognitive-behavioural intervention originally developed for use in pharmacotherapy trials for AUD and has demonstrated feasibility and acceptability in similar populations. The intervention content draws on established CBT strategies for alcohol reduction, including motivational enhancement, managing triggers, coping skills, and relapse prevention.
  Other Names: Take Control Cognitive Behavioural Therapy Module
Other: Placebo — Participants in the placebo condition will receive visually-matched sham injections, where by the placebo container and contents will be identical in appearance to Tirzepatide, except without the active ingrediant.
  Arms: Placebo: subcutaneous administration of placebo plus CBT ("Take Control" program)

SUMMARY:
The investigators approach is to conduct a Phase II Double-Blind randomised controlled trial with individuals with co-occurring Alcohol Use Disorder and overweight/obesity (AUD-OOB) to receive either a sub-cutaneous injection of Tirzepatide (2.5 mg for 4 weeks followed by 5 mg for 4 weeks) or visually matched sham saline injection, in combination with a structured behavioural intervention (Take Control CBT Module). The primary aim of the study is evaluate the efficacy of the intervention on the number of heavy drinking days (defined as 5+ standard drinks for men, 4+ standard drinks for women) during the final month of treatment (weeks 5 to 8) compared to baseline. The secondary aim of the study is to assess treatment effects on alcohol related (e.g. number drinks consumed per day, abstinent days) and cardio-metabolic outcomes (e.g. body weight in kg, waist circumference, blood pressure, HbA1c, total cholesterol etc...), and summarise safety outcomes associated with use (e.g. frequency and severity of side effects, number of serious adverse events, treatment related discontinuations). The study will also include neurobiological assessments such as functional magnetic resonance imaging (fMRI) and lab-based psychophysiology to assess the impact of tirzepatide on change in brain activity and autonomic responses to alcohol and food cues.

DETAILED DESCRIPTION:
Individuals with co-occurring AUD and overweight or obesity (AUD-OOB) are an underserved population with high relapse rates and elevated cardiometabolic risk. Recent evidence suggests that Tirzepatide can simultaneously reduce alcohol intake in animal models and craving, drinks per day and heaving drinking days over a 9-week period in non-treatment seeking individuals with AUD. Tirzepatide's dual incretin mechanism offers the potential to simultaneously reduce alcohol use and improve metabolic health in this group, with a favourable safety profile and weekly dosing that supports adherence. As rates of AUD and obesity continue to rise, identifying pharmacological strategies that can address both conditions concurrently is a high public health priority.

This is a phase II, randomised, double-blind, placebo-controlled clinical trial of 46 individuals designed to evaluate the effects of Tirzepatide on alcohol consumption, craving and cardiometabolic outcomes in adults with alcohol used disorder and overweight/obesity (AUD-OOB), to receive either a sub-cutaneous injection of tirzepatide (n=23) or a visually matched placebo (n=23).

The trial will be conducted at a single clinical site in New South Wales, Australia. The Edith Collins Centre (ECC) will serve as the coordinating centre.

In summary participants will:

* Be randomized in a double-blind fashion to receive either tirzepatide or a visually matched placebo
* Receive subcutaneous injections of tirzepatide (2.5mg for 4 weeks followed by 5mg for 4 weeks) or a matching placebo over an eight-week treatment period.
* Visit the clinic weekly (for 8 weeks) for medication administration, clinical monitoring and brief behavioural support (delivered by the "Take Control" computerised CBT program).
* Receive clinical assessments including alcohol use, cardiometabolic biomarkers (HbA1c, lipids, ASCVD) and alcohol biomarkers (PEth) at baseline (week 0), end of treatment (week 9) and follow-up (week 12).
* Undergo neuroimaging (fMRI) and psychophysiology assessmenrts as a substudy at 2 timepoints: baseline (week 0) and between week 7-9. These tasks will assess neural and autonomic reactivity to alcohol and food-related cues, and will support a mechanistic understanding of tirzepatide's impact on reward sensitivity and stress responsivity-key predictors of relapse and treatment outcome

The primary aim of this clinical trial is to examine the effects of weekly tirzepatide (2.5 mg for 4 weeks followed by 5 mg for 4 weeks) versus placebo injections, in combination with a structured behavioural intervention (Take Control) on alcohol consumption in adults with alcohol use disorder and overweight/obesity (AUD-OOB). The main question[s] it aims to answer are:

1. Main outcome: To determine the efficacy of Tirzepatide on alcohol related outcomes, the change in the number of heavy drinking days during the final four weeks of treatment (week 5 - 8, with a final assessment at week 9) will be assessed by comparison with baseline (28 days prior to baseline visit). Researchers will compare tirzepatide to placebo injections (a look-alike substance that contains no drug) to see if weekly tirzepatide administration can reduce the number of heavy drinking days.
2. Secondary Outcomes:

   i) To evaluate changes in additional alcohol-related outcomes:
   * Number of drinks per drinking day measured using the Timeline Follow Back
   * Number of abstinent days measured using the Timeline Follow Back
   * WHO drinking risk level
   * Weekly alcohol craving
   * Proportion of participants with zero heavy drinking days (Weeks 5-8)

   ii) To evaluate changes in cardiometabolic indices from baseline to Week 9:
   * Body weight
   * Waist circumference
   * Blood pressure
   * HbA1c
   * Total cholesterol
   * Triglycerides
   * 10-year ASCVD risk score

   iii) To assess safety outcomes associated the delivery of Tirzepatide, investigators will measure the:
   * Frequency and severity of side effects (graded using CTCAE V5.0 and monitored continuously throughout the intervention).
   * Number of serious adverse events (SAEs)
   * Treatment-related discontinuation

   Participants will complete additional neurobiological assessments including functional magnetic resonance imaging (fMRI) and laboratory-based psychophysiology at two timepoints: baseline (pre-treatment) and the final treatment visit (Week 8), which coincides with the final tirzepatide/placebo dose and final Take Control session. These measures will assess changes in brain activity and autonomic responses to alcohol and food cues.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 to 75 years
2. Meet DSM-5 criteria for alcohol use disorder (AUD) with at least moderate severity (≥4 symptoms in the past year)
3. Have an average daily alcohol consumption of:

   * ≥60g ethanol/day for men
   * ≥40g ethanol/day for women (based on the 28 days prior to the baseline visit)
4. Body mass index (BMI) ≥27 kg/m²
5. Currently motivated to reduce or stop drinking but not engaged in formal AUD treatment
6. Able and willing to attend weekly clinic visits and complete all study procedures
7. Fluent in English and able to provide informed consent
8. Stable housing situation (not transient or homeless)

Exclusion Criteria:

1. Past-year DSM-5 diagnosis of another substance use disorder (except nicotine or mild cannabis use disorder)
2. Recent (past 30 days) self-reported illicit drug use (excluding cannabis), or a positive urine drug screen for non-cannabis substances
3. History of significant alcohol withdrawal, defined by:

   * History of seizure, delirium tremens, or
   * Hospitalisation for withdrawal, or
   * CIWA-Ar score >9, or
   * PAWS score >4 at screening
4. Currently engaged in pharmacological or behavioral treatment for AUD, or prior engagement within the past 3 months
5. History or current diagnosis of:

   * Type 1 or Type 2 diabetes
   * Diabetic complications (e.g. retinopathy)
   * HbA1c ≥6.5% at screening
6. Significant psychiatric illness, including:

   * Current active suicidal ideation (per C-SSRS)
   * Lifetime history of psychosis or bipolar disorder
   * Unstable depression or anxiety interfering with daily functioning
7. Chronic or acute pancreatitis
8. Significant liver disease or abnormal liver function tests (ALT, AST, ALP, bilirubin >3× ULN)
9. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) type I/II
10. Estimated glomerular filtration rate (eGFR) <30 mL/min
11. Recent significant weight loss (>5% of body weight in past 30 days)
12. Use of any weight loss medication (e.g., orlistat, bupropion-naltrexone) or AUD medication (e.g., naltrexone, acamprosate, topiramate, varenicline) in the past 3 months
13. Use of tirzepatide or any GLP-1 receptor agonist in the past 6 months
14. Pregnant or breastfeeding, or not using effective contraception (females of childbearing potential)
15. Inability to attend weekly visits due to work/travel/schedule conflicts
16. Participation in another clinical trial involving an investigational product
17. Shared household with a current or past participant in this trial
18. Scheduled for surgery requiring anaesthesia within 90 days of enrolment that would interfere with participation or follow-up
19. History of muscle wasting, bone disorders (e.g. sarcopenia)
20. Active gastrointestinal conditions that could interfere with treatment (e.g., severe GERD)
21. Uncontrolled hypertension, recent heart attack or stroke (within 6 months)

    Extra Exclusion criteria for Those Participants Agreeing to Participate in Neuroimaging & Psychophysiology Tasks:
22. Presence of any MRI-incompatible metal implants or devices, including pacemakers, aneurysm clips, insulin pumps, or cochlear implants
23. History of brain surgery or penetrating head trauma
24. Prior occupation as a machinist, welder, or metal worker (due to risk of metal fragments)
25. Non-removable piercings or dental hardware that would interfere with MRI
26. History of claustrophobia likely to interfere with scanning compliance aa. Neurological disorders (e.g., epilepsy, multiple sclerosis) likely to confound neuroimaging data bb. Inability to lie still or tolerate MRI procedures cc. Patient weighting over 159kg (MRI scan limit) dd. Any other condition or medication judged by the investigator to preclude safe participation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Heavy Drinking Days | 12 weeks (measured at baseline, during the final 4 weeks of treatment [weeks 5 - 8], end of treatment [week 9], and follow-up [week 12]).
  Reduction in Heavy Drinking Days (HDD; defined as 4 or more drinks in a day for women and 5 or more drinks in a day for men). This will be measured by the Timeline Follow Back.

SECONDARY OUTCOMES:
Number of drinks per drinking day consumed | 12 weeks (weekly, from baseline visit to final follow-up visit at week 12)
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
Abstinent days | 12 weeks (weekly, from baseline visit to final follow-up visit at week 12)
  Measured by Timeline Follow Back
Alcohol Craving | 12 weeks (weekly, from baseline visit to final follow-up visit at week 12)
  As measured the Visual Analogue Scale (VAS) weekly and also at pre-, during-, and post- psychophysiological cue-reactivity task completion. Scored from to 0 to 100, where higher scores indicate more severe craving.
WHO drinking risk level scale. | 12 weeks (weekly, from baseline visit to final follow-up visit at week 12)
  The WHO drinking risk level scale categorizes alcohol consumption based on average daily intake of pure alcohol (in grams) and its associated health risk.
  There are 5 levels that differ based on gender:
  * For men, very high risk >100 grams/day or; high risk as >60 to 100 grams/day ; moderate risk as >40 to 60 grams/day; and low risk as 1 to 40 grams/day.
  * For women, very high risk was defined as >60 grams/day; high risk as >40 to 60 grams/day; moderate risk as >20 to 40 grams/day ; and low risk as 1 to 20 grams/day.
Proportion of participants with zero heavy drinking days | 4 weeks (weeks 5 to 8)
  Proportion of participants with zero heavy drinking days measured by the TLFB.
Body weight | Measured at baseline [week 0] and at end of treatment [week 9].
  Changes in body weight in kilograms (kg) from baseline to week 9 (end of treatment).
Waist circumference | Measured at baseline [week 0] and at end of treatment [week 9]
  Changes in waist circumference in centimetres (cm) from baseline to week 9 (end of treatment).
Blood pressure | 9 weeks (weekly, from baseline visit to final dose at week 8)
  Systolic and diastolic blood pressure measured weekly from baseline to end of treatment (week 8).
HbA1c | 3 weeks (Measured at baseline [week 0] and at end of treatment [week 9], and week 12 if clinically indicated)
  Clinical metabolic monitoring for cardiometabolic risk and drug safety. Measures glycated haemoglobin in a blood in percentages (%). Collected at screening (Week 0) and again at the end-of-treatment visit (Week 9). Additional testing may be conducted at follow up (week 12) if clinically indicated.
10-year ASCVD risk score | Measured at baseline [week 0] and end of treatment [week 9].
  A cardiometabolic biomarker providing an estimation of 10-year atherosclerotic cardiovascular disease (ASCVD) risk score, based on pooled cohort equations. This is a composite risk score derived from traditional cardiovascular risk factors, including gender, age, race, total cholesterol, total HDL cholesterol, systolic BP, previous receipt of treatment for high blood pressure (if SBP > 120 mmHg), diabetes and smoking status.
  This is used to provide a risk score of atherosclerotic cardiovascular disease.
Frequency and severity of side effects/adverse events (AEs) | 12 weeks (at each visit)
  Safety outcomes including adverse events (AEs), serious adverse events (SAEs), and vital sign abnormalities, will be summarised descriptively across the study period. Feasibility outcomes (e.g., recruitment and retention rates, session attendance) will be analysed using proportions with corresponding 95% confidence intervals.
Number of treatment-related discontinuation | 12 weeks (at each visit)
  As a measure of safety, the number of treatment-related discontinuations will be measured.
Total cholesterol | 3 weeks (Measured at baseline [week 0] and at end of treatment [week 9], and week 12 if clinically indicated)
  Clinical metabolic monitoring for total cholesterol in millimoles per litre (mmol/L). Collected at screening (Week 0) and again at the end-of-treatment visit (Week 9). Additional testing may be conducted at follow up (week 12) if clinically indicated.
Triglycerides | 3 weeks (Measured at baseline [week 0] and at end of treatment [week 9], and week 12 if clinically indicated)
  Clinical metabolic monitoring for triglycerides in blood sample, measured via millimoles per litre (mmol/L) as a measure of cardiometabolic risk and drug safety. Collected at screening (Week 0) and again at the end-of-treatment visit (Week 9). Additional testing may be conducted at follow up (week 12) if clinically indicated.
Changes in Positive and Negative Mood States | Week 1 (prior to dose 1) and at EOT (end of treatment/week 8)
  Mood states before/after ketamine sessions assessed by PANAS (Positive and Negative Affect Schedule). This will be measured during neuroimaging and psychophysiology sessions. Used to measure an individual's emotional state, assessing two dimensions: Positive Affect (PA; captures feelings like enthusiasm and alertness), and Negative Affect (NA; measures distress and negative emotions like anger and anxiety).
Alcohol craving measure 2 | 12 weeks - measured weekly from baseline (week 1) to outcomes/discharge (week 12)
  As measured by the Penn Alcohol Craving Scale (PACS). 5-item self-report questionnaire that evaluates alcohol craving over the past week. Measures frequency, intensity, duration of craving, perceived control over drinking, and overall craving severity. Each item is rated on a 7-point Likert scale (0-6). Total scores range from 0 to 30, with higher scores indicating greater craving.

OTHER OUTCOMES:
Changes in cigarette use | At baseline (week 0) and at end-of-treatment visit (week 9).
  Measured according to the average number of cigarettes smoked per day, only among participants who reported regular smoking at baseline. Analysed with a mixed-effects models.
Changes in cannabis use | At baseline (week 0) and at end-of-treatment visit (week 9).
  Measured according to the average number of days of cannabis used per week, only among participants who reported baseline use. Analysed with a mixed-effects models.
Changes in phosphatidylethanol (PEth), an objective biomarker of alcohol use | Baseline (Week 0), End-of-treatment (week 9) and optionally at week 12
  Changes in PEth (phosphatidylethanol) from baseline to Week 9 will be analysed using MMRM, with baseline PEth as a covariate. Collected at week 0, 9 (end-of-treatment) and optionally at week 12.
Changes in depressive symptom severity | At baseline (week 0) and at end-of-treatment visit (week 9).
  Measured by cumulative scores on the Center for Epidemiologic Studies Depression Scale (CES-D). This scale consists of 20 items with a minimum score of 0 and a maximum score of 60. A higher score indicates greater depressive symptomatology. Items are rated according to how often the feeling or behavior occurred in the past week (e.g. 0 = Rarely or none of the time (less than 1 day; 1 = Some or a little of the time (1-2 days); 2 = Occasionally or a moderate amount of the time (3-4 days) and 3 = Most or all of the time (5-7 days))
Change in sleep disturbance and sleep problems | At baseline (week 0) and at end-of-treatment visit (week 9).
  As measured by cumulative scores Insomnia Severity Index (ISI). This scale consists of 7 items with a minimum total score of 0 and a maximum score of 28. A higher score indicates greater insomnia severity. Items are rated on a 0-4 scale based on the severity or impact of sleep difficulties over the past two weeks (e.g., 0 = No problem; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very severe).
  A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "sub-threshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)."
Change in health-related quality of life | At baseline (week 0) and at end-of-treatment visit (week 9).
  As measured by cumulative scores on the 36-Item Short Form Health Survey (SF-36). Consists of 36 items grouped into 8 domains of health:
  1. Physical Functioning (10 items)
  2. Role Limitations due to Physical Health (4 items)
  3. Role Limitations due to Emotional Problems (3 items)
  4. Energy/Fatigue (4 items)
  5. Emotional Well-being (5 items)
  6. Social Functioning (2 items)
  7. Pain (2 items)
  8. General Health (5 items)
  Each item is scored from 0 to 100, with higher scores indicating better health status. Items are rated based on experiences over the past 4 weeks using Likert-type response options (e.g., ranging from "All of the time" to "None of the time" or "Excellent" to "Poor").
  Items within a domain are summed and averaged, then transformed to a 0-100 scale. Refer to the following reference for specific transformations needed for each item: https://www.rand.org/health/surveys/mos/36-item-short-form/scoring.html
Daily fluctuations in alcohol use, craving, and mood | Daily throughout the 12 weeks using the SEMA application
  Measured through the use of Ecological Momentary Assessment (SEMA) via smartphone prompts.
Evaluation of treatment acceptability | Week 9 and optional Week 12
  Collected via structured post-treatment feedback at Week 9 and optional qualitative interviews at Week 12.
Alcohol urge | Week 0 and Week 9 (before and after the Psychophysiological cue-reactivity tasks [if agreed to by the participant])
  To assess short term alcohol urge, the Alcohol Urge Questionnaire (AUQ) will be used. This is a brief 8-item self-report questionnaire that evaluates acute alcohol craving as a single factor (unidimensional). Each item is rated on a Likert scale of 7 points, with higher scores indicating stronger urges to consume alcohol. Two of the questions are reversed scored.
Changes in anxiety symptom severity | At baseline (week 0) and at end-of-treatment visit (week 9).
  Measured by cumulative scores on the GAD-7 (Generalised Anxiety Disorder 7-item scale). Measures anxiety symptom severity over the last two weeks, and the extent to which the participant is bothered by these symptoms.
  Each item is scored from 0 to 3 (where 0 = not at all, 1= several days, 2= more than half of days, 3=nearly every day). This scale has a minimum score of 0 and a maximum score of 21. A higher score indicates greater severity of generalized anxiety symptoms (The total score indicates anxiety severity: 0-4 is minimal anxiety, 5-9 is mild, 10-14 is moderate, and 15-21 is severe).
Changes in suicidal ideation using the Columbia Suicide Severity Rating Scale (C-SSRS). | 12 weeks (measured weekly)
  The C-SSRS is a structured clinician-administered instrument with strong predictive validity for suicidal behavior, used in clinical and research settings to assess the presence, severity, and intensity of suicidal ideation and behavior. The C-SSRS is administered by trained clinicians. C-SSRS scoring includes four subscales: ideation severity (items 1-5, scored by the most severe type endorsed); intensity of ideation (sum of five items including frequency, duration, controllability, deterrents, and reasons for ideation; range 2-25; higher number indicates more intense ideation); suicidal behavior (presence or absence of actual, interrupted, aborted, or preparatory behavior recorded separately); and potential lethality (medical damage rated 0-5, potential lethality rated 0-2). At baseline, this is measured by the baseline version. Higher scores indicate more severe suicidality.
Withdrawal Status | Prior to neuroimaging at baseline [week 0] and the final imaging date [between week 7 and 9].
  To determine changes in the severity of alcohol withdrawal symptoms the Revised Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar) will be used. This 10-item scale evaluates common withdrawal symptoms including nausea/vomiting, tremor, paroxysmal sweats, anxiety, agitation, tactile disturbances, auditory disturbances, visual disturbances, headache and orientation. Each item is rated on a scale from 0 to 7 (except orientation, which is rated 0-4), with a total score ranging from 0 to 67. Higher scores indicate more severe withdrawal symptoms.
Depression severity | Measured weekly from baseline (week 1) to outcomes/discharge (week 12)
  As measured by the Patient Health Questionnaire-9 (PHQ-9). A 9-item self-report instrument that assesses the severity of depressive symptoms over the past two weeks. Items correspond to DSM-5 criteria for major depressive disorder, including mood, interest, sleep, energy, appetite, self-worth, concentration, psychomotor changes, and suicidal thoughts. Each item is rated on a 4-point Likert scale (0 = "Not at all" to 3 = "Nearly every day"). Total scores range from 0 to 27, with higher scores indicating greater depressive symptom severity.
Changes in withdrawal status (#2) | Measured weekly from baseline (week 1) to final follow up visit (week 12)
  As measured by the Short Alcohol Withdrawal Scale (SAWS). A self-report questionnaire designed to assess the severity of alcohol withdrawal symptoms over the past 24 hours. It consists of 10 items covering common withdrawal symptoms such as anxiety, tremor, sweating, nausea, sleep disturbance, and sensory sensitivity. Each item is rated on a 4-point Likert scale (0 = "Not at all" to 3 = "Severe"). Total scores range from 0 to 30, with higher scores indicating greater withdrawal severity.
To determine risk of severe alcohol withdrawal | Measured at screening (first visit) to determine withdrawal severity status
  As measured by the Prediction of Alcohol Withdrawal Severity Scale (PAWSS). A clinician-administered screening tool designed to predict the risk of developing severe alcohol withdrawal complications (e.g., seizures, delirium tremens) in patients. Consists of 10 items which assess recent alcohol use, history of withdrawal complications, and clinical risk factors (e.g., elevated blood alcohol level, concurrent use of sedatives). Each item is scored as 0 (absent) or 1 (present). Total scores range from 0 to 10, with higher scores indicating greater risk. A score of ≥4 suggests high risk for severe withdrawal.
Alcohol use severity | Measured at baseline
  As measured by the Alcohol Use Disorders Identification Test (AUDIT). A 10-item screening questionnaire used to identify hazardous and harmful alcohol consumption, as well as possible alcohol dependence. Items cover three domains:
  1. Alcohol consumption (frequency, quantity, binge drinking)
  2. Alcohol-related problems (injury, guilt, concern from others)
  3. Dependence symptoms (impaired control, morning drinking)
  Each item is scored from 0 to 4, giving a total score range of 0-40, with higher scores indicating greater risk. Common interpretation thresholds:
  0-7: Low risk 8-12: Risky drinking 13+: High risk
Nicotine dependence | Measured at baseline
  As measured by the Fagerström Test of Nicotine Dependence (FTND). A 6-item self-report questionnaire which assess the intensity of physical addiction to nicotine. Items evaluate behaviors such as time to first cigarette after waking, daily cigarette consumption, difficulty refraining from smoking in forbidden places, and smoking patterns during the day. Each item is scored on a scale (0-1 or 0-3 depending on the question), with a total score range of 0-10, where higher scores indicate greater nicotine dependence.
  Common interpretation thresholds:
  0-2: Very low dependence 3-4: Low dependence 5: Medium dependence 6-7: High dependence 8-10: Very high dependence
Impulsive traits | Measured at baseline
  As measured by the UPPS Impulsive Behavior Scale. This is a self-report questionnaire designed to assess multidimensional impulsivity across five distinct facets:
  1. Negative Urgency (acting rashly under distress)
  2. Positive Urgency (acting rashly under extreme positive emotions)
  3. Lack of Premeditation (difficulty thinking before acting)
  4. Lack of Perseverance (difficulty staying focused on tasks)
  5. Sensation Seeking (tendency to seek excitement and novel experiences) This version contains 59 items. Responses are rated on a Likert scale (typically 1 = "Strongly agree" to 4 = "Strongly disagree"). Scores are calculated for each facet, with higher scores indicating greater impulsivity in that domain.
Difficulty controlling alcohol consumption | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by the Impaired Control Scale (ICS). A self-report questionnaire which assesses difficulty in controlling alcohol consumption. It includes items evaluating perceived inability to stop drinking once started, failure to adhere to drinking limits, and loss of control over drinking behavior. Responses are typically rated on a Likert scale, with higher scores indicating greater impaired control.
Measure of positive reinforcement from the environment | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by the Environmental Reward Observation Scale (EROS). A self-report measure assessing the degree to which individuals experience positive reinforcement from their environment, and evaluates engagement in rewarding activities and perceived availability of environmental rewards. Items are rated on a Likert scale, with higher scores indicating greater environmental reinforcement.
Drinking frequency in high-risk situations | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by a multi-item questionnaire titled Inventory of Drinking Situation scale. This scale assesses high-risk situations for drinking, such as coping with negative emotions, social pressure, and positive mood states. Responses indicate frequency or likelihood of drinking in these contexts. Higher scores suggest greater vulnerability to relapse.
Reward driven eating tendencies | Measured weekly from baseline (week 1) to final follow up visit (week 12)
  As measured by the Reward-Based Eating Drive Scale (R-BEDS). A self-report tool assessing compulsive eating behaviors driven by reward sensitivity. It evaluates loss of control over eating, lack of satiety, and preoccupation with food. It consists of 9 items, each rated on a Likert scale from 1 to 5:
  * 1 = Strongly Disagree
  * 5 = Strongly Agree
  Items are grouped into three subscales:
  1. Loss of Control Over Eating
  2. Lack of Satiety
  3. Preoccupation With Food
  Total Scores range from 9 to 45, where higher scores indicate greater reward-driven eating tendencies.
Presence and severity of food addiction symptoms | Measured at baseline
  As measured by the Yale Food Addiction Scale (YFAS). Assesses addictive-like eating behaviors based on DSM criteria for substance use disorders. It measures symptoms such as tolerance, withdrawal, loss of control, and continued use despite negative consequences. Scoring identifies 1) symptom count ranging from 0 to 7 reflecting number of addiction like criteria endorsed with higher scores indicating greater food addiction severity; and 2) a dichotomous "diagnosis" that indicates whether a threshold of 3/< "symptoms" plus clinically significant impairment or distress is satisfied.
Trait level food craving tendencies | Measured at baseline and at follow-up 1 (safety outcomes, week 9)
  Measured by the General Food Craving Questionnaire - Trait (G-FCQ-T). This is a self-report measure that assesses the general tendency to experience food cravings over time. It includes multiple subscales. Items are rated on a Likert scale, with higher scores indicating stronger trait-level food cravings. There are 21 items scored on a Likert scale ranging from 1 = never to 6 = always, with a score range between 21 and 126. Higher scores are indicative of more frequent and intense trait food cravings.
Anhedonia (ability to experience pleasure in last few days) | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by the Snaith-Hamilton Pleasure Scale (SHPS). A self-report questionnaire which assesses anhedonia across domains such as social interactions, food and drink, sensory experiences, and hobbies. Items are rated on a Likert scale, with the final score ranging from 14 to 56. Higher scores indicate greater anhedonia. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree.
Self-efficacy for maintaining abstinence | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by the Alcohol Abstinence Self-Efficacy Scale (AASE). Self report measure assessing confidence in resisting alcohol use across high-risk situations (e.g., negative emotions, social pressure). Items are rated on a Likert scale, with higher scores indicating greater self-efficacy for maintaining abstinence. Each item is scored on a scale from 1 (not at all confident) to 5 (extremely confident) relating to the level of confidence a participant has to not drink alcohol.
Compulsions and obsessive thoughts related to alcohol use | Measured at baseline (week 1), dosing visit 5 (mid-point of medication schedule) and at the first (safety outcome, week 9) and second follow-up visits (outcomes/discharge, week 12)
  As measured by the Obsessive-Compulsive Drinking Scale (OCDS). A 14-item questionnaire that measures an individual's severity of obsessive thoughts and compulsions to use alcohol. Includes two subscales 1. obsessions (thoughts, urges) and 2. compulsions (drinking behaviors). Higher scores indicate greater cognitive and behavioral preoccupation with alcohol. Each item is scored on a scale of 0 to 4.
Food cravings at a specific point in time | Measured weekly from baseline (week 1) to final follow up visit (week 12)
  As measured by the General Food Craving Questionnaire-State (G-FCQ-S). A self-report measure assessing momentary food cravings at a specific point in time. Items capture craving intensity, desire, and preoccupation. Higher scores indicate stronger state-level cravings.
Intensity of cigarette craving | Measured weekly from baseline (week 1) to final follow up visit (week 12)
  As measured by the Tiffany Questionnaire of Smoking Urges (QSU). Measures the intensity and nature of cigarette craving, assessing 2 dimensions:
  1. Desire and intention to smoke for positive reinforcement (e.g., pleasure, satisfaction) and....
  2. Urgency to smoke to relieve negative affect or withdrawal symptoms There are 32 items, each rated on a 7-point Likert scale ranging from 1= strongly disagree to 7 = strongly agree. Higher total summed scores are indicative of a stronger craving and motivation to smoke.
Motivation and demand for alcohol. | Measured weekly from baseline (week 1) to final follow up visit (week 12)
  As measured by the Alcohol Purchase Task (APT). Measure assesses demand and motivation for alcohol under varying price conditions. Participants indicate how many drinks they would purchase at different prices. Outcomes include indices such as intensity, elasticity, and breakpoint, reflecting motivation and valuation of alcohol.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haber, MD, RACP, FAChAM, Principal Investigator — Sydney Local Health District
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No